CLINICAL TRIAL: NCT00221819
Title: Prospective Study of the Influence of the Humidification Mode on Ventilation Parameters and Arterial Blood Gases in Non Invasive Ventilation
Brief Title: Gases Humidification During Noninvasive Ventilation : Heat and Moisture Exchanger or Heated Humidifier ?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 9300-02
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2013-05

CONDITIONS: Acute Lung Injury; Pneumonia; Chronic Obstructive Pulmonary Disease; Acute Heart Failure
Keywords: Humidification; Heat and moisture exchanger; Heated humidifier, non invasive ventilation
MeSH Terms: conditions — Acute Lung Injury; Pneumonia; Pulmonary Disease, Chronic Obstructive

INTERVENTIONS:
Device: heated humidifier (device)
Device: Heat and moisture exchanger (device)

SUMMARY:
To humidify gases during non invasive ventilation, both to heated humidifier (HH) and heat and moisture exchanger (HME) are routinely used. Patients receiving non invasive ventilation for acute respiratory failure were randomized to HME or HH. The purpose of this study was to evaluate respiratory parameters and arterial blood gases (ABG) of patients during NIV with small dead space HME compared to HH.

DETAILED DESCRIPTION:
Objective: Few data are reported in the field of noninvasive ventilation (NIV) regarding humidification devices. It was previously suggested that standard heat and moisture exchangers (HME) had adverse gasometrical and clinical outcomes in acute respiratory failure (ARF) of chronic respiratory failure patients (CRF). This study was performed to evaluate respiratory parameters and arterial blood gases (ABG) of patients during NIV with small dead space HME compared to heated humidifier (HH).

Design: Prospective randomized cross-over study. Setting: A 16-bed medical intensive care unit (ICU) and a 14-bed medico surgical ICU.

Patients: Patients receiving NIV for ARF in the context of CRF or hypoxic ARF and patients with persistent weaning failure receiving NIV just after extubation.

Measurements: HME and HH were randomly compared during 2 NIV periods of 30 minutes separated by a 20 to 30 minutes period of spontaneous breathing with oxygen. ABG were collected at baseline and at the end of each period. As well as respiratory parameters including volumes, pressures, P0.1, a comfort score, capnometry and oxygen saturation. Two sets of patients were successively studied whether they have a flex tube added to the ventilatory circuit or not.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving NIV for ARF in the context of CRF, hypoxic ARF or patients with persistent weaning failure receiving NIV just after extubation

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-06; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Air blood gases at the end of each study period (one with HME, one with HH)

SECONDARY OUTCOMES:
Respiratory parameters including volumes, pressures, P0.1, a comfort score, capnometry and oxygen saturation at the end of each study period (one with HME, one with HH)

CONTACTS AND LOCATIONS:
Overall Officials: alexandre Boyer, Dr, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Département de Réanimation Médicale, Hôpital Pellegrin-Tripode, Place A. Raba Léon,, Bordeaux, France